CLINICAL TRIAL: NCT01602861
Title: The Effects of Spironolactone on Calcineurin Inhibitor Induced Nephrotoxicity
Acronym: SPIREN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Fredericia Hosptial (Other)
Responsible Party: Principal Investigator, Line Aas Mortensen, Principal Investigator, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Eudra CT: 2011-002243-98
Record Dates: First submitted 2012-05-17; First posted 2012-05-21 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Disorder Related to Renal Transplantation
Keywords: Fibrosis; calcineurin inhibitor; kidney transplant; chronic rejection
MeSH Terms: conditions — Fibrosis | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spironolactone (Experimental)
  Interventions: Drug: Spironolactone
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Spironolactone — One tablet per day (25 mg Spironolactone/placebo) for the first three months. Subsequently dosage is increased to two tablets per day (50 mg Spironolactone/placebo) for the rest of the study.
  In case of hyperkaliemia (>5,5 mmol/L) or intolerable side effects dosage will be reduced to one tablet per day (25 mg Spironolactone/placebo).
  Arms: Spironolactone
Drug: placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess whether the diuretic drug spironolactone can prevent chronic damage to transplanted kidneys caused by the medication that prevents rejection.

Spironolactone prevents the effects of the hormone aldosterone. Aldosterone is suspected of being involved in the processes leading to chronic rejection of transplanted kidneys. Hence, by blocking the effects of aldosterone we hope to be able to prevent loss of kidney function in transplant patients.

DETAILED DESCRIPTION:
AIM: The purpose of this study is to assess whether spironolactone can prevent the formation of fibrosis in transplanted kidneys.

BACKGROUND: Calcineurin inhibitors (CNI) are one of the cornerstones of immunosuppressive therapy after kidney transplantation. The introduction of CNI has caused a significant decrease in acute rejections. However, CNI also have known side effects. These include the formation of tubulointerstitial fibrosis in the transplanted kidney, contributing over time to impaired kidney function and reduced graft survival.

The mineralocorticoid aldosterone may be involved in the development of renal fibrosis. Recent observations suggest that aldosterone plays a central role in the pathogenesis of CNI nephrotoxicity and that the mineralocorticoid-receptor-blocker spironolactone could be a useful agent to prevent it.

METHODS: This study is a randomized, placebo-controlled, double-blind study in which 170 renal transplant patients will be recruited from two nephrological departments in Southern Denmark. Patients will be randomized to three years of treatment with either spironolactone or placebo added to the standard immunosuppressive treatment. Renal graft biopsies, various molecular tests of tissue, blood and urine, chrome-EDTA clearance, 24-hour bloodpressure measurement and blood samples will be performed at inclusion, after 1 year, 2 years and upon completion.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Proteinuria < 3 g/24 hours
3. Creatinine clearance ≥ 30 mL/min
4. S-Potassium < 5,5 mmol/L
5. Negative pregnancy test at the inclusion and anticonception

Exclusion Criteria:

1. Intolerance to spironolactone
2. Creatinine clearance < 30 ml/min
3. S-Potassium ≥ 5,5 mmol/L
4. Resin or digoxine treatment
5. Pregnancy or planned pregnancy
6. Relevant organic, systemic or mental illness
7. Anticipation of lack of compliance or understanding the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2013-02; Primary Completion 2021-04 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Change in Cr EDTA clearance | 0, 1 year, 2 years, 3 years

SECONDARY OUTCOMES:
Reduced urine protein levels (change from baseline) | 0, 1 year, 2 years, 3 years
Reduced fibrosis (change from baseline) | 0, 2 years
  Verified by graft biopsies and immuno histochemistry. Newly transplanted patients will be subjected to additional biopsies 3 months and 1 year after inclusion.
Reduced blood pressure (change from baseline) | 0, 1 year, 2 years, 3 years
Cardiovascular events | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Claus Bistrup, MD, ph.d., Study Director — Dep. of Nephrology, Odense University Hospital
Locations (1):
- Odense University Hospital, Odense C, Denmark

REFERENCES:
- [Derived] Natale P, Mooi PK, Palmer SC, Cross NB, Cooper TE, Webster AC, Masson P, Craig JC, Strippoli GF. Antihypertensive treatment for kidney transplant recipients. Cochrane Database Syst Rev. 2024 Jul 31;7(7):CD003598. doi: 10.1002/14651858.CD003598.pub3. PMID 39082471
- [Derived] Mortensen LA, Thiesson HC, Tougaard B, Egfjord M, Fischer ASL, Bistrup C. The effect of spironolactone on calcineurin inhibitor induced nephrotoxicity: a multicenter randomized, double-blind, clinical trial (the SPIREN trial). BMC Nephrol. 2018 May 3;19(1):105. doi: 10.1186/s12882-018-0885-6. PMID 29724188